CLINICAL TRIAL: NCT01296230
Title: Varicocelectomy: Can Sex-hormones Predict Improvements in Semen Quality?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to recruit participants
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-2-2010-067
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2012-02

CONDITIONS: Varicocele; Infertility; Semen Quality
MeSH Terms: conditions — Varicocele; Infertility | interventions — Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hormone/semen measurements before and after varicocelectomy (Experimental): We will measure sex-hormone and semen quality in patients both before and after varicocelectomy. The purpose is to asses if preoperative hormone levels are predictive for who will have improved semen quality after surgery.
  Interventions: Procedure: Hormone and semen measurements before varicocelectomy

INTERVENTIONS:
Procedure: Hormone and semen measurements before varicocelectomy — Before surgery we will measure sex-hormone levels and semen parameters. This will be repeated after the varicocelectomy to record any changes.

SUMMARY:
The purpose of this study is to determine if the pre-operative levels of sex-hormones can be used to identify the varicocele patients who can expect improvements in their semen parameters following varicocelectomy.

ELIGIBILITY:
Inclusion Criteria:

* Varicocele (grade 1-3) and surgery planned for this condition
* At least 18 years of age

Exclusion Criteria:

* Fever within 3 months before the first semen sample
* Malformations of the uro-genital tract
* Karyotype other than 46, XY or Y micro deletions
* Endocrine disease
* Chronic disease
* Medications which reduce semen quality
* Epididymitis within 6 months before surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Change in semen parameters | February 2017 (anticipated duration of the study)

SECONDARY OUTCOMES:
Change in hormone levels | February 2017 (anticipated end of the study)

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - University Department of Growth and Reproduction GR, Section 5064, Rigshospitalet, Copenhagen
  - Department of Urology, Herlev Hospital, Herlev